CLINICAL TRIAL: NCT05775094
Title: A Pilot Study of Romosozumab Efficacy and Safety for the Management of Myelomarelated OsteoLytic Disease in Postmenopausal Women With Multiple Myeloma and Osteoporosis (REMOLD-MM)
Brief Title: A Study of Romosozumab in Women With Multiple Myeloma and Osteoporosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-038
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Osteoporosis; Multiple Myeloma
Keywords: Romosozumab; 23-038
MeSH Terms: conditions — Osteoporosis; Multiple Myeloma | interventions — romosozumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Romosozumab (Experimental): Romosozumab will be given on-label for osteoporosis at 210 mg administered SC once monthly for 12 months in conjunction with antimyeloma therapy.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Romosozumab will be administered 210 mg SC as two 105 mg prefilled syringes once every 4 weeks x 12 months. No dose adjustments for romosozumab will be permitted. All efforts will be made to administer romosozumab within the defined study visit windows (+/- 14 days).

SUMMARY:
The purpose of this study is to measure the effect of romosozumab on bone formation and breakdown (resorption) and determine if romosozumab is a safe treatment for osteoporosis and myeloma-related bone disease (MBD) in postmenopausal people with multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Documented MM per International Myeloma Working Group diagnostic criteria (evidence of myeloma defining event attributed to underlying plasma cell disorder): i. Clonal plasma cells in the bone marrow ≥ 10% or presence of a biopsy proven plasmacytoma; and ii. Any one or more of the following myeloma defining events:
* Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder:

  1. Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11 mg/dL)
  2. Renal insufficiency: creatinine clearance < 40 mL/min or serum creatinine 177µmol/L (>2 mg/dL)
  3. Anemia: hemoglobin > 2 g/dL below the lower limit of normal, or a hemoglobin value <10 g/dL
  4. Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET/CT
* Clonal bone marrow plasma cell percentage ≥ 60%; or
* Involved: uninvolved serum free light chain (FLC) ratio ≥ 100 (involved FLC level be ≥ 10 mg/dL; or
* >1 focal lesion on MRI studies (at least 5 mm in size)
* Presence of lytic bone lesion(s) due to MM based on radiographic evidence with at least one measurable lesion (≥0.5 cm in its largest diameter by computerized tomography [CT])
* Postmenopausal female, defined as last menstrual cycle at least 12 months prior to study enrollment
* Must have one of the following:

  * osteoporosis on dual X-ray absorptiometry (DXA) scan; or
  * fragility fracture of the spine or hip; or
  * morphometric spine fracture; or
  * osteopenia with elevated risk of fracture (calculated by the FRAX online calculator)
* Within 12 months prior to study entry, ≤ 4 doses of prior intravenous (IV) bisphosphonate with the last dose ≥ 3 months prior to study entry.
* Prior oral bisphosphonates are allowed if the last dose was ≥ 3 months prior to study entry.
* Prior denosumab use is allowed for the following:

  * For patients who received ≤ 5 consecutive doses of denosumab with the last dose of denosumab received ≥ 3 months prior to study entry.
  * For patients who received ≥ 6 doses of denosumab, IV bisphosphonate should be given at least 1 month after the last dose of denosumab (if the last dose of denosumab was within the past 2 years). Patients are then eligible ≥ 3 months after IV bisphosphonate is received. If ≤ 2 years have elapsed since the last dose of denosumab, IV bisphosphonate is not required, and patients are eligible for the study.
* Signed informed consent form(s). Individuals with impaired decision-making capacity may enroll if legally authorized representatives consent on behalf of individuals with impaired decision-making capacity.
* Ability to comply with all study-related procedures in the investigator's judgment
* 18 years of age or older

Exclusion Criteria:

* Assigned male at birth
* Received teriparatide or other PTH analog use within 12 months prior to study entry
* Receiving concurrent antiresorptive therapy
* History of cardiovascular event (myocardial infarction and/or stroke) within the past 12 months of study entry
* History of non-healed dental or oral surgery
* History of osteonecrosis of the jaw
* 25 (OH) vitamin D levels < 20 ng/mL. Vitamin D repletion will be permitted and subjects may be rescreened once 25 (OH) vitamin D level ≥ 20 ng/mL.
* Current hyper- or hypocalcemia, defined as albumin-adjusted serum calcium outside the normal range per institutional standard (<8.5 or >10.5 mg/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women are at high risk for fractures.
Enrollment: 10 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percent change in bone formation marker, P1NP | up to 2 years

SECONDARY OUTCOMES:
Incidence and severity of adverse events | up to 2 years
  evaluating adverse events using NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Carlyn Tan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm